CLINICAL TRIAL: NCT07042087
Title: Lifestyle for the BRAin Health - Time Restricted Eating and Mindfulness
Acronym: LIBRA REMIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Slovak Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16V/2024; 101087124 (Other Grant/Funding Number: Horizon EU)
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Aging; Lifestyle Factors; Cognitive Impairment; Yoga; Time Restricted Eating; Diet Modification
Keywords: Alzheimer's Disease Prevention; Mindfulness-Based Intervention; Cognitive Training; Time-Restricted Eating; Dietary consultation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Intermittent Fasting | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Yoga and Time-Restricted Eating Intervention (Experimental): Participants in this arm will take part in a 9-month intervention consisting of yoga-based mindfulness sessions combined with time-restricted eating (16:8 protocol). The yoga program includes physical postures (asanas), breathing techniques, and meditation, aimed at improving physical fitness, stress regulation, and cognitive function. The dietary component promotes a flexitarian diet within an 8-hour daily eating window. Sessions are conducted twice weekly for 90 minutes under certified instructors.
  Interventions: Behavioral: Mindfulness Yoga; Behavioral: Time-Restricted Eating with nutritional counseling promoting a flexitarian dietary pattern
- Cognitive Training and Stretching Intervention (Active Comparator): Participants in this arm will engage in a 9-month intervention including cognitive training exercises and guided stretching. The cognitive program targets multiple domains: verbal and non-verbal memory, executive functions, attention, language, and social cognition. Sessions are delivered twice weekly for 90 minutes by trained therapists. This intervention serves as an active comparator for assessing the effects of yoga and dietary modification on cognitive and biological outcomes.
  Interventions: Behavioral: Cognitive Training; Behavioral: Stretching

INTERVENTIONS:
Behavioral: Mindfulness Yoga — A structured 9-month program integrating physical yoga postures (asanas), breathing techniques, sound, and meditation. Sessions are conducted twice weekly (90 minutes each) and focus on enhancing physical health, stress regulation, and cognitive performance. Delivered by certified instructors.
  Arms: Mindfulness Yoga and Time-Restricted Eating Intervention
Behavioral: Time-Restricted Eating with nutritional counseling promoting a flexitarian dietary pattern — Participants follow a 16:8 time-restricted eating schedule (16 hours fasting / 8 hours eating window) for 9 months, with nutritional counseling promoting a flexitarian dietary pattern. The intervention is designed to support metabolic health and reduce risk factors for neurodegeneration.
  Arms: Mindfulness Yoga and Time-Restricted Eating Intervention
Behavioral: Cognitive Training — A 9-month structured program of twice-weekly cognitive training sessions (90 minutes each), targeting memory, attention, executive function, and social cognition using both paper-based and computer-based tasks. Supervised by trained therapists.
  Arms: Cognitive Training and Stretching Intervention
Behavioral: Stretching — A twice-weekly stretching routine performed over 9 months (90-minute sessions), led by physiotherapists. This intervention provides low-intensity physical activity to control for physical engagement across study arms.
  Arms: Cognitive Training and Stretching Intervention

SUMMARY:
The study aims to evaluate the effects of a 9-month intervention combining yoga-based mindfulness techniques, cognitive training, and nutritional counseling on cognitive function, plasma markers of neurodegeneration (tau protein), physical fitness, and metabolism in older adults at increased risk of developing Alzheimer's disease.

DETAILED DESCRIPTION:
This randomized two-arm clinical trial aims to evaluate the effects of a 9-month intervention combining yoga-based mindfulness techniques and time-restricted eating (Arm 1) versus cognitive training and stretching (Arm 2) in older adults at increased risk of developing Alzheimer's disease. The study will assess outcomes including cognitive function, plasma biomarkers of neurodegeneration (tau protein), physical fitness, and metabolic health.

The trial is harmonized with the concurrently running LIBRA-NET study (NCT06986096) conducted at Slovak sites (Bratislava and Banská Bystrica). Data from the cognitive training arm and additional clinical parameters will be pooled across both studies for joint statistical analyses. The studies share primary and several secondary outcomes, a shared intervention timeline, assessment protocols, and the cognitive training/stretching arm. The harmonization across all four study sites aims to increase statistical power and enable more generalizable conclusions for a larger population.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 years
* Diagnosis of Subjective Cognitive Impairment (SCI) or Mild Cognitive Impairment (MCI)
* mini-mental-scale (MMSE) score between 24-30
* Positive plasma pTau217 biomarker
* Stable dose of iAChE therapy (if applicable)
* Ability to participate in a 9-month intervention

Exclusion Criteria:

* Stroke or myocardial infarction within the past year
* Decompensated internal conditions (e.g., severe heart failure, kidney failure, unstable diabetes, GLP1 agonist therapy)
* Long-term psychiatric treatment (except well-managed depression)
* Neurological conditions affecting mobility or cognition (e.g., Parkinson's disease, severe tremor, epilepsy)
* Severe sensory or motor impairment preventing protocol participation
* Active cancer treated within the past 5 years
* Poor anticipated compliance (e.g., transport issues, time constraints, non-cooperation)
* Concurrent participation in another clinical study
* Unstable iAChE medication regimen
* Substance or alcohol dependence

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite Score of Cognitive Function | Baseline and 9 months
  Change in composite neuropsychological score from baseline to post-intervention (9 months), including domain-specific scores for memory, executive function/attention, and psychomotor speed.
Plasma Biomarkers of Neurodegeneration | Baseline and 9 months
  Change in concentrations of plasma biomarkers: phosphorylated tau (pTau217, pTau181), GFAP, and neurofilament light chain (NfL).

SECONDARY OUTCOMES:
Computerized Cognitive Test Scores - Cogstate | Baseline and 9 months
  Change in individual and composite scores on computerized cognitive tests (e.g., Cogstate), including measures of spatial orientation.
Geriatric depression scale | Baseline and 9 months
  Changes in depression, using the GDS scale
Adherence to Intervention | Throughout the 9-month intervention
  Attendance rate and adherence to prescribed intervention protocol (minimum attendance threshold and dietary compliance).
Beck's anxiety inventory | Baseline and 9 months
  Anxiety levels measured by the BAI
Older People's Quality of Life Questionnaire scores | Time Frame: Baseline and 9 months
  Quality of life measured by OPQOL-35

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Sheardova, MD. PhD., Principal Investigator — The International Clinical Research Center of St. Anne's University Hospital in Brno (FNUSA-ICRC)
Locations (1):
- Fnusa/ Icrc, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No